CLINICAL TRIAL: NCT02290327
Title: Re-Evaluating the Inhibition of Stress Erosions: Gastrointestinal Bleeding Prophylaxis In ICU
Acronym: REVISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REV-06MAR14
Record Dates: First submitted 2014-10-31; First posted 2014-11-14 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-02

CONDITIONS: Stress Ulcer Prophylaxis
Keywords: Stress ulcer bleeding; proton pump inhibitors; pneumonia; clostridium difficile infection
MeSH Terms: conditions — Pneumonia; Clostridium Infections | interventions — Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 50 ml of 0.9% Normal Saline Intravenously once daily
  Interventions: Drug: Placebo
- Pantoprazole (Active Comparator): Pantoprazole 40 mg in 50 ml 0.9% Normal Saline Intravenously once daily
  Interventions: Drug: Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole — Proton pump inhibitor
  Arms: Pantoprazole
Drug: Placebo — 50 ml of 0.9% normal saline
  Arms: Placebo

SUMMARY:
The purpose of the this Pilot Trial is to determine the feasibility of conducting a large randomized controlled trial (RCT), that aims to examine the efficacy and safety of using pantoprazole compared to placebo for stress ulcer prophylaxis in critically ill mechanically ventilated patients in the ICU.

DETAILED DESCRIPTION:
Background For almost 4 decades, stress ulcer prophylaxis to prevent upper gastrointestinal (GI) bleeding has been standard of care in the ICU. The 1999 American Society of Health-System Pharmacists guidelines recommend stress ulcer prophylaxis for the critically ill. The 2013 Surviving Sepsis Campaign guidelines recommend stress ulcer prophylaxis for patients mechanically ventilated for > 48 hours or with coagulopathy. However, GI bleeding rates are significantly lower today than in the past, potentially reduced by optimal resuscitation and early enteral nutrition. Additional concerns include whether acid suppression has any impact on bleeding at all, and whether acid suppression does more harm than good, given the apparent increased risk of more common, serious problems of pneumonia and Clostridium difficile infection. Further, prophylaxis has become almost universal rather than targetted at patients at risk of GI bleeding. Thus, clinicians and investigators globally are calling for a re-evaluation of acid suppression with a large Randomized controlled trial (RCT) comparing proton pump inhibitor against placebo.

Objectives To determine the feasibility of performing a large RCT to investigate whether intravenously administered pantoprazole, compared to placebo prevents clinically important gastrointestinal bleeding in mechanically ventilated patients in the intensive care unit (ICU), based on 3 outcomes: the informed consent rate; recruitment rate, and protocol adherence

Design Prospective, concealed, stratified, randomized, blinded, multicentre trial.

Setting Canadian and Saudi medical-surgical university-affiliated ICUs.

Methods Patients will be stratified by center, and medical/surgical/trauma status, then will be randomized to intervention or placebo using an allocation ratio of 1:1 and undisclosed variable block sizes. Research pharmacists will prepare identical 100ml mini-bags of the pantoprazole 40mg or placebo with blinded research labels for once daily dosing.

Followup Research Coordinators in the ICU will review all patients daily, where most of the trial data will be collected. This will involve baseline data (e.g., demographics, illness severity, advanced life support), and daily data (e.g., study medication administered and reasons why not administered), other relevant medications and co-interventions that might influence bleeding, ventilator associated pneumonia (VAP) or Clostridium difficile outcomes (e.g., enteral nutrition, antibiotics, anticoagulants, possible VAP prevention strategies including probiotics), laboratory, microbiology, transfusion or radiology documentation to help adjudicate the outcomes of clinically important and overt bleeding, VAP, and Clostridium difficile infection, and mortality. We do not anticipate any loss to follow up; we expect to have complete follow up of patients in the ICU.

Patients will be followed for primary and secondary outcomes during their ICU stay on daily basis. Once patients are discharged from the ICU, they will no longer be followed daily; only duration of hospital stay and vital status at hospital discharge will be obtained.

A secure web-based central randomization method will ensure site-specific stratified allocation tables. When the patient is identified as eligible and consent is obtained by Research Coordinator, the Research Pharmacist will take the assignment and dispense study drug accordingly.

Relevance Results of the REVISE Pilot Trial will provide key feasibility and safety data which will serve to plan a larger multicentre trial of pantoprazole versus placebo for stress ulcer prophylaxis in mechanically ventilated critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years
2. Anticipated invasive mechanical ventilation of ≥48 hours, determined by the intensivist

Exclusion Criteria:

1. Invasive mechanical ventilation >72 hours before randomization.
2. Patients who must receive PPI due to active bleeding or increased bleeding risk (e.g., patients with acute GI bleeding, recent severe esophagitis, Zollinger Ellison syndrome, Barrett's esophagus, peptic ulcer bleeding within 8 weeks [mild dyspepsia or mild gastroesophageal reflex disease will not be excluded])
3. Receiving dual antiplatelet therapy aspirin and clopidogrel prior to randomization
4. Palliative care or decision to withdraw advanced life support (patients with a decision to forgo cardiopulmonary resuscitation will not be excluded)
5. Previous enrolment in this or a related trial
6. Pregnancy
7. Physician, patient, or substitute decision maker (SDM) declines
8. Two or more 'daily doses' of prophylaxis with H2RA or PPI (one day of a single PPI dose is not an exclusion criterion if once daily dosing of PPI prophylaxis was administered; one day of bid [twice daily] dosing of an H2RA is not an exclusion criterion if twice daily H2RA prophylaxis was administered; one day of tid [thrice daily] dosing of an H2RA is not an exclusion criterion if thrice daily H2RA prophylaxis was administered).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Consent Rate | 12 months
  This will be calculated as the overall proportion of consented patients of those substitute decision makers (SDMs) approached (with 95% CI).
  A successful consent rate will be defined as ≥70% of SDMs approached to consent.
Recruitment Rate | 12 months
  A successful recruitment rate will be defined as achieving enrolment of 90 patients, conventionally expressed as 2 patients per center per month over 12 months.
Protocol Adherence | 12 months
  This will be calculated as doses of study drug administered as a proportion of doses prescribed and associated 95% confidence intervals.
  A successful adherence will be defined as ≥80% of prescribed drugs being administered.

SECONDARY OUTCOMES:
Clinically important upper gastrointestinal bleeding | During ICU stay (expected average is 10 days)
Ventilator associated pneumonia | During ICU stay (expected average is 10 days)
Mortality | During ICU and hospital stay (expected average ICU stay is 10 days, expected average hospital stay is 30 days)
Clostridium Difficile infection | During ICU stay (expected average ICU stay is 10 days)

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Alhazzani, MD,FRCPC,MSc, Principal Investigator — McMaster University
Locations (10):
- Royal Adelaide, Adelaide, Australia
- Canada (8):
  - Queen Elizabeth II, Halifax, Nova Scotia
  - St. Joseph's HealthCare Hospital, Hamilton, Ontario
  - Jurvinski Hospital, Hamilton, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Ottawa Civic Hospital, Ottawa, Ontario
  - Ottawa General Hospital, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - St Michael's Hospital, Toronto, Ontario
- Dammam University, Dammam, Eastern Province, Saudi Arabia

REFERENCES:
- [Derived] Alhazzani W, Guyatt G, Marshall JC, Hall R, Muscedere J, Lauzier F, Thabane L, Alshahrani M, English SW, Arabi YM, Deane AM, Karachi T, Rochwerg B, Finfer S, Daneman N, Zytaruk N, Heel-Ansdell D, Cook D, Of OB. Re-evaluating the Inhibition of Stress Erosions (REVISE): a protocol for pilot randomized controlled trial. Ann Saudi Med. 2016 Nov-Dec;36(6):427-433. doi: 10.5144/0256-4947.2016.427. PMID 27920416